CLINICAL TRIAL: NCT03466632
Title: Randomised Study Comparing the Use of Propofol Versus the Use of Dexmedetomidine as a Sedative Agent for Patients Presented for Lower Gastrointestinal Endoscopy
Brief Title: Propofol Versus the Use of Dexmedetomidine as a Sedative Agent for Colonosopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dexmedetomidine colonoscopy
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Propofol Group (Active Comparator): propofol 1.5 mg/kg slow intravenously, followed by maintenance dose of 0.5 mg/kg/h throughout the procedure..
  Interventions: Drug: Propofol
- • Dexmedetomidine Group (Active Comparator): dexmedetomidine 1 ug/kg over 10 minutes as a bolus dose followed by continuous infusion at a dose of 0.5 ug/kg/h as maintenance dose throughout the procedure
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — propofol 1.5 mg/kg slow intravenously, followed by maintenance dose of 0.5 mg/kg/h throughout the procedure.
  Arms: • Propofol Group
Drug: Dexmedetomidine — dexmedetomidine 1 ug/kg over 10 minutes as a bolus dose followed by continuous infusion at a dose of 0.5 ug/kg/h as maintenance dose throughout the procedure
  Arms: • Dexmedetomidine Group

SUMMARY:
Dexmedetomidine as a Sedative Agent for Patients Presented for Lower Gastrointestinal Endoscopy

DETAILED DESCRIPTION:
Propofol Versus the Use of Dexmedetomidine as a Sedative Agent for Patients Presented for Lower Gastrointestinal Endoscopy

ELIGIBILITY:
Inclusion Criteria:

* aged 25-45 years,
* ASA class I or II,
* who are scheduled for elective outpatient colonoscopy

Exclusion Criteria:

* refused to give informed consent
* if they had known hypersensitivity to the used drugs
* patients with morbidly obese patients
* patients with increased risk for airway obstruction as obstructive sleep apnea,
* Liver diseases

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adequate sedation | 6 months
  the number of patients adequately sedated

CONTACTS AND LOCATIONS:
Overall Officials: Sherief Abd-Elsalam, MD, Study Director — Tanta University; Sameh Abdelkhalek Ahmed, MD, Study Director — Tanta University Anasthesia Department
Locations (1):
- Sameh Abdelkhalek Ahmed, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided